CLINICAL TRIAL: NCT01199133
Title: A Randomised,Double-blind,Placebo-controlled,Multi National,Phase III Trial to Assess the Efficacy and Safety of 300 IR Sublingual Immunotherapy Administered as Allergen-based Tablets Once Daily to Adolescents and Children Above the Age of 5 Years, Suffering From House Dust Mite Allergic Rhinitis
Brief Title: Safety and Efficacy Study of Sublingual Immunotherapy (SLIT) to Treat House Dust Mite Allergic Rhinitis in Adolescents and Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study population was insufficiently symptomatic to enable evaluation of the efficacy of the treatment. No safety concern.
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VO64.08; 2009-011999-30 (EudraCT Number)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Allergic Rhinitis Due to Dust Mite
MeSH Terms: interventions — Allergens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 300 IR (Active Comparator): 300 IR house dust mites allergen extract tablet
  Interventions: Drug: 300 IR house dust mites allergen extract tablet
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 300 IR house dust mites allergen extract tablet — One sublingual tablet daily for one year.
  Other Names: House dust mites (Der p and Der f) allergen extract tablet
  Arms: 300 IR
Drug: Placebo tablet — One sublingual tablet daily for one year.
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of one dose of sublingual immunotherapy (SLIT) administered to children and adolescents as allergen-based tablets once daily over a period of 24 months over 3 years compared to placebo, for reduction of allergic rhinitis symptoms and rescue medication use.

DETAILED DESCRIPTION:
After the screening period, the patients will be administered 300 IR house dust mite allergen based tablets or placebo, once a day, for a period of 36 months with two windows of 8 months and 6 months without treatment. The carry over effect will be evaluated after a treatment free follow up period of 24 months.

An independent Data Monitoring Committee will be constituted to evaluate the efficacy and safety data at the end of Year 1 and Year 3, and the post-treatment long-term efficacy data at the end of year 4.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, aged 5-17 years inclusive
* History of house dust mite-related allergic rhinitis for at least 1 year requiring regular intake of symptomatic treatment(s)
* Sensitised to D. pteronyssinus and/or D. farinae (positive skin prick test with wheal diameter greater than 3 mm and specific IgE level ≥ 0.7 kU/L)

Exclusion Criteria:

• Co-sensitization associated with clinically relevant allergic rhinitis, sinusitis, conjunctivitis or asthma likely to significantly change the symptoms of the patient throughout the study (that means patient symptomatic to another allergen than house dust mites to which the patient will be exposed during the study, i.e. will notably be excluded

* patients sensitised to cat or dog allergens and regularly exposed to these allergens
* patients sensitised to aspergillus, cladosporium, alternaria
* patients sensitised to parietaria , ragweed, or mugwort, if this allergen is endemic to the region

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 471 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Wahn, MD, Study Chair — Charite- Campus Virchow klinikum

REFERENCES:
- [Derived] Worm M, Demoly P, Okamoto Y, Vidal C, Daghildjian K, Yan K, Casale TB, Bergmann KC. Safety of 300IR house dust mite sublingual tablet from pooled clinical trial and post-marketing data. World Allergy Organ J. 2024 Jun 25;17(7):100924. doi: 10.1016/j.waojou.2024.100924. eCollection 2024 Jul. PMID 39035788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 27 OCT 2009, Last Patient Last Visit 30 SEP 2011
Period: Year 1
Arm/Group | 300 IR | Placebo
Started | 241 | 230
Completed | 211 | 215
Not Completed | 30 | 15
Not completed — Adverse Event | 16 | 4
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Any other reason not above-mentioned | 6 | 7
Period: Year 2
Arm/Group | 300 IR | Placebo
Started | 211 | 215
Completed | 208 | 212
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Any other reason not above-mentioned | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all randomized patients who received at least one dose of study treatment and had at least one evaluation of Adjusted Symptom Score (AdSS) during the treatment Year 1 period.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR | Placebo | Total
Number analyzed (Participants) | 222 | 221 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.0 (3.24) | 11.2 (3.41) | 11.1 (3.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 81 | 156
  Male | 147 | 140 | 287

OUTCOME MEASURES:

1. Primary Outcome: Average Adjusted Symptom Score (AASS) During the Treatment Period
Description: The primary efficacy endpoint was the Average Adjusted Symptom Score (AAdSS) during the period from 1 October 2010 to 30 November 2010 (Year 1 Primary Period) assessed in the Full Analysis Set defined for Year 1. The Average Adjusted Symptom Score (AAdSS) ranges from 0 to 12, with a higher score meaning a worse outcome.
  It is a score assessing four rhinitis symptoms: sneezing, rhinorrhoea, nasal pruritus and nasal congestion, adjusted on the rescue medication intake
Time Frame: Year 1 Primary Period = 01 OCT to 30 NOV 2010 The value was obtained by averaging the daily scores over the primary period
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 222 | 221
units on a scale | 2.85 (0.160) | 2.84 (0.155)
Statistical Analysis 1: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA; Difference in LS Means = 0.01, 95% CI [-0.41 to 0.43]

ADVERSE EVENTS:
Time Frame: Reporting and collection of Adverse Events go from the date of the first administration of investigational product up to the 30th day (inclusive) after the last administration in Year 1 treatment period, a total of 13 months.
Description: Treatment Emergent Adverse Event (TEAE) defined as any Adverse Event which started on or after the date of the first administration of investigational product up to the 30th day (inclusive) after the last administration in Year 1 treatment period.
  A treatment Emergent Adverse Event is not necessarily a treatment related adverse event. "Treatment Emergent" refers to temporality, not to causality.
Arm/Group | 300 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 8/241 | 7/230
Other Adverse Events (participants affected / at risk) | 149/241 | 124/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=241) | Placebo (N=230)
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Varicocele (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=241) | Placebo (N=230)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 36
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 | 30
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 24 | 6
Pharyngitis (Infections and infestations) | 23 | 21
Bronchitis (Infections and infestations) | 22 | 28
Tonsillitis (Infections and infestations) | 14 | 4
Upper respiratory tract infection (Infections and infestations) | 13 | 9
Nasopharyngitis (Infections and infestations) | 10 | 15
Oral pruritus (Gastrointestinal disorders) | 27 | 7
Abdominal pain (Gastrointestinal disorders) | 14 | 4
Tooth loss (Gastrointestinal disorders) | 13 | 8
Tongue oedema (Gastrointestinal disorders) | 13 | 0
Headache (Nervous system disorders) | 21 | 23
Pyrexia (General disorders) | 5 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No